CLINICAL TRIAL: NCT05543291
Title: Multi-omics Analysis of Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ai Peng, Shanghai tenth People's Hospital, Shanghai 10th People's Hospital
Other Study IDs: SHYS-IEC-5.0/22K162/P01
Record Dates: First submitted 2022-09-11; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Potential Mechanisms Underlying the Microbiota-Gut-Kidney Axis in CKD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal and serum samples were collected for metagenome and metabolome analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy controls
  Interventions: Behavioral: renal function
- mild CKD
  Interventions: Behavioral: renal function
- Moderate CKD
  Interventions: Behavioral: renal function
- ESRD
  Interventions: Behavioral: renal function

INTERVENTIONS:
Behavioral: renal function — levels of eGFR

SUMMARY:
Chronic kidney disease (CKD) is a progressive disease with hidden epidemics and one of the most significant contributing factors to end-stage renal disease (ESRD), cardiovascular comorbidities, cachexia and anemia, which accounts for a nearly 1.2 million populations died per year.

ELIGIBILITY:
Inclusion Criteria:

Age-matched and gender-matched HC with normal renal and liver function and not taking any medications were enrolled

Exclusion Criteria:

1. Age<18 years.
2. Individuals with hypertension, diabetes, obesity, metabolic syndrome or pregnancy.
3. Individuals who received gastrointestinal operation, antibiotics or probiotic products within one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  1. Confirmed CKD patients.
  2. Age≥18 years.
  Exclusion criteria：
  1. Age<18 years.
  2. Patients with active gastrointestinal diseases, liver cirrhosis, cancer, active infection or cardiovascular event in the past 3 months, pregnancy or received renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional and structural alteration of microbiotas and their crosstalk with CKD-associated metabolism | baseline
  Gut metagenome, fecal metabolome and serum metabolome were performed in this disease-severity classified CKD cohort, to identify the changes of microbial compositions and metabolism in CKD progression

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrolgoy, Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang H, Xue W, Cheng J, He Y, Song Y, Hu D, Peng A, Li C, Bao H. Altered fecal microbial and metabolic profiles reveal potential mechanisms underlying anemia in patients with chronic renal failure. Microbiol Spectr. 2025 Aug 5;13(8):e0316624. doi: 10.1128/spectrum.03166-24. Epub 2025 Jun 17. PMID 40525868